CLINICAL TRIAL: NCT06177951
Title: Improving the Transition to Home for Moderate to Late Preterm Infants Admitted to the NICU Through Parent Education and Discharge Preparation
Brief Title: Using NICU Discharge Education Tools to Enhance Discharge Preparation for Parents of Moderate to Late Preterm Infants
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 23-0490
Record Dates: First submitted 2023-12-11; First posted 2023-12-20 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Discharge Readiness

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control Group (No Intervention): This group will receive neither of the interventions (NICU Discharge Passport, NICU Infant Care Class).
- Received NICU Discharge Passport Only (Experimental): This group will receive only one intervention: NICU Discharge Passport.
  Interventions: Other: NICU Discharge Passport
- Received NICU Infant Care Class Only (Experimental): This group will receive only one intervention: NICU Infant Care Class.
  Interventions: Other: NICU Infant Care Class
- Received Both NICU Discharge Passport and NICU Infant Care Class (Experimental): This group will receive both interventions: NICU Discharge Passport, NICU Infant Care Class.
  Interventions: Other: NICU Discharge Passport; Other: NICU Infant Care Class

INTERVENTIONS:
Other: NICU Discharge Passport — The NICU discharge passport contains a discharge checklist highlighting important "go-to" information for infants (feeding plan, medications, pharmacy information, pediatrician, and follow ups post-discharge). It also provides key anticipatory guidance for newborns.
  Arms: Received Both NICU Discharge Passport and NICU Infant Care Class; Received NICU Discharge Passport Only
Other: NICU Infant Care Class — The class will be provided once or twice weekly to eligible study participants. It will be conducted in a small group format. Class teachers will focus on providing key anticipatory guidance to aid in the transition home during the first month of life . Topics related to infant care will be discussed, including feeding, elimination, skincare, hygiene, soothing, development, and when to see a doctor/emergencies.
  Arms: Received Both NICU Discharge Passport and NICU Infant Care Class; Received NICU Infant Care Class Only

SUMMARY:
The goal of this clinical trial is to improve the transition to home for preterm infants born between 33-36 weeks gestational age and discharged from the neonatal intensive care unit (NICU) through the use of two interventions, a "NICU Discharge Passport" and "NICU Infant Care Class," for parents.

The main question[s] the clinical trial aims to answer are the impact of the above discharge interventions on:

* parental readiness for discharge
* feasibility of compliance with discharge instructions
* number of ER/urgent visits and hospital re-admission rates 1-month post-discharge

Participants will include parents/guardians and nurses of eligible preterm infants discharged from the Cohen Children's Medical Center NICU. Baseline data will be collected for a period of 4-6 months for a control group (who will receive current NICU discharge practices), after which two interventions will be implemented for a period of 4-6 months to the intervention groups. Interventions will include: a) NICU Discharge Passport and b) NICU Infant Care Class.

Data collection will include pre and post-discharge surveys for parent and nurse participants in charge of discharging the eligible infant participant. Surveys will assess parental readiness for discharge, compliance with discharge instructions, ER/urgent visits post-discharge, hospital re-admission rates post-discharge, and if applicable, obtain feedback on interventions.

Researchers will compare responses between control and intervention groups to understand the impact of the interventions on parental discharge preparedness.

DETAILED DESCRIPTION:
Currently, parents of 33-36 weeks gestational age neonates discharged from the NICU receive discharge-related information, including feeding plan, medications, follow up appointments, and more, from their discharge summary completed in the electronic medical record. This moderate to late preterm population is a unique transitory preterm population in the NICU because while these infants do not face the same risk of medical complications as their younger counterparts, they do require more focused management for very specific risks of prematurity, including poor oromotor skills, glycemic control, thermoregulation, and immature development. Furthermore, much of their short admission period in the NICU is spent in both the management of these concerns and the provision of parental education and support for the same.

The objective of this study is to improve the transition to home for 33-36 weeks gestational age preterm infants discharged from the NICU through the use of a specific "NICU Discharge Passport" and "NICU Infant Care Class" for parents. The study hypothesis is that these interventions will improve parental discharge preparedness.

Study participants will include parents/guardians and nurses of eligible preterm infants discharged from the Cohen Children's Medical Center NICU. Baseline data will be collected for a period of 4-6 months for a control group (who will receive current NICU discharge practices), after which two interventions will be implemented for a period of 4-6 months to the intervention groups. Interventions will include: a) NICU Discharge Passport, consisting of a discharge checklist and key anticipatory guidance for newborns and b) NICU Infant Care Class, provided in person weekly to all eligible study participants.

Data collection will include surveys for parents and nurses. Parents will complete a total of 2 surveys (one before discharge from the hospital, the second at a 1-month follow up survey via telephone). Nurses will complete 1 survey before discharge of the infant participant from the NICU. Survey details: The pre-discharge survey will be administered to both parents and nurses, and assess parental readiness for discharge home with their child. In addition, for parents receiving the interventions, the pre-discharge survey will obtain feedback regarding the interventions. The pre-discharge survey will be completed within the 5-day period leading up to discharge once the infant is identified by the medical team as a discharge candidate. One month post discharge from the hospital, a follow up phone call survey will be obtained from all parents participating in the study. The post-discharge survey will again assess parental readiness for discharge home with their child. It will also collect information on parental self-report on the transition home from the NICU, including any barriers encountered. Researchers will compare survey responses between control and intervention groups.

ELIGIBILITY:
Inclusion Criteria:

* Parent and/or legal guardian of all preterm infants born at a gestational age (GA) between 33 weeks and 0 days, and 36 weeks and 6 days, at Cohen Children's Medical Center (CCMC) that will be admitted to and discharged from the NICU will be included in this study.
* A maximum of one parent/guardian for each eligible infant will be included in the study.
* Twin infants will be treated as separate study subjects.
* The nurse in charge of discharging the eligible infant will be included in the study.

Exclusion Criteria:

* Parents of infants not being discharged to home from CCMC NICU (ie discharged to rehab and/or other facilities).
* NICU patients with a diagnosis of congenital heart disease requiring intervention during current admission (This is due to the fact that these patients already have specific discharge instructions/transition plan(s) in place).
* Parents/guardians that are Non-English speaking will be excluded from the study due to the inability of the current study to provide all interventions in non-English languages.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2024-01-08 (Actual); Primary Completion 2024-09-08 (Estimated); Study Completion 2024-10-08 (Estimated)

PRIMARY OUTCOMES:
Parental Readiness for Hospital Discharge | Pre-discharge, 1-month Post-discharge
  Parental readiness for discharge will be assessed through survey questions administered to both nurse and parent participants. Parent participants will answer the questions pre-discharge and 1-month post-discharge. Nurse participants will answer the questions pre-discharge. The survey will consist of 10 questions on a Likert scale (responses are assigned numerical points which will be summed to obtain a readiness score). The questions will assess parental confidence, preparation, knowledge, and support at home in regards to discharge with their infant.

SECONDARY OUTCOMES:
Number of ER/Urgent Visits | 1-month Post-Discharge
  At follow up survey, 1-month post-discharge from the hospital, parent participants will be asked how many ER and/or urgent visits they have had since leaving the NICU.
Hospital Re-admission Rates | 1-month Post-Discharge
  At follow up survey, 1-month post-discharge from the hospital, parent participants will be asked if their child has required re-admission since discharge from the NICU.
Adherence to Discharge Instructions | 1-month Post-Discharge
  At follow up survey, 1-month post-discharge from the hospital, parent participants will be asked how feasible it has been to follow their baby's discharge plan, including feeding instructions, practicing safe sleep, administering medications, and following up with their pediatrician.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Sullivan, MD, Principal Investigator — ksullivan14@northwell.edu
Locations (1):
- Cohen Children's Medical Center, Queens, New York, United States

IPD SHARING:
Plan to Share IPD: No